CLINICAL TRIAL: NCT03786627
Title: The Effect of Combined Neuromuscular Electrical Stimulation and Motor Control Training on Lumbar Multifidus Muscle Activation in Individuals With Impaired Lumbopelvic Control
Brief Title: Neuromuscular Electrical Stimulation and Motor Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Principal investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/199.1010
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Instability; Back
Keywords: Clinical lumbar instability; History of low back pain; Arthrogenic muscle inhibition; Neuromuscular electrical stimulation; Motor control training

STUDY DESIGN:
Intervention Model Description: Subjects with impaired lumbopelvic control will be randomly assigned to either combined NMES with motor control training group, or motor control training alone group using randomly generated number in concealed envelopes.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Physical therapist, investigator, and assessor will be blinded to the group assignment. This process will be handled by the research coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined NMES and motor control (Experimental): This group will receive combined 15-minute neuromuscular electrical stimulation and 30-minute motor control training based on movement system impairment concept.
  Interventions: Other: Combined NMES and motor control
- Motor control and placebo NMES (Placebo Comparator): This group will receive placebo NMES for 15 minutes followed by 30 minutes motor control training based on movement system impairment concept.
  Interventions: Other: Motor control and placebo NMES

INTERVENTIONS:
Other: Combined NMES and motor control — This group will receive the neuromuscular electrical stimulation using interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect) on bilateral lumbar multifidus muscles. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total stimulation time is 15 minutes. After that, this group will receive 30 minutes motor control training. This motor control training will focus on the control of the lumbar multifidus muscle in various functional tasks. It is believed to restore the motor units in individuals with arthrogenic muscle inhibition. This motor control training will take approximately 30 minutes. This group will receive intervention twice a week for 8 weeks.
  Arms: Combined NMES and motor control
Other: Motor control and placebo NMES — This group will the neuromuscular electrical stimulation without turning the electrical current for 15 minutes. After that, this group will receive 30 minutes motor control training. This motor control training will focus on the control of the lumbar multifidus muscle in various functional tasks. This motor control training will take approximately 30 minutes. This group will receive intervention twice a week for 8 weeks.
  Arms: Motor control and placebo NMES

SUMMARY:
Phase I, this study aims to:-

1. Establish intra- and inter-rater reliability and minimal detectable change of ultrasound imaging measurement
2. Determine appropriate mode and dose for neuromuscular electrical stimulation on lumbar multifidus muscle
3. Determine feasibility of proposed protocol and physical therapy intervention

Phase II, this study aims to:-

1. Determine the difference lumbar multifidus muscle activation based on arthrogenic muscle inhibition model between individuals with and without impaired lumbopelvic control
2. Determine the effect of combined neuromuscular electrical stimulation and motor control training in individual with impaired lumbopelvic control

DETAILED DESCRIPTION:
Phase I: Preliminary study Subjects aged between 20 and 40 with and without history of low back pain will be recruited. Subjects who are interested in participation will undergo a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If they meet all inclusion criteria, the consent process will be performed.

After obtaining the written informed consent, all subjects will fill out the information sheet for demographic data. The body landmarks will be identified. These landmarks include 1) lumbar spinous process of L2-L5, 2) L4-5 facet joint (2 cm lateral to inferior one half of spinous process of L4), and 3) lumbar multifidus muscle (2 cm lateral to L5 spinous process and 3 cm lateral to L2 spinous process). Bilateral L4-5 facet joints will be used to place ultrasound transducer for capturing lumbar multifidus muscle, while location of lumbar multifidus muscle will be used to place NMES electrodes. Then, subjects will undergo clinical outcome measures including clinical observation of aberrant movement pattern during functional movements, passive SLR, hamstrings muscle length test, modified Thomas's and Ober's tests, abdominal and back muscle strength.

The subjects will be in prone position on treatment table with thorax (T3 level) and pelvis (S2 level) securely fastened to the bed. Hand-held dynamometer will be placed at the thorax to measure back extension force. Then, ultrasound transducer will be placed at right L4-5 facet joint by rater-A. Right lumbar multifidus muscle activation at rest will be recorded. Then, rater-A will move the transducer to left L4-5 facet joint to measure left lumbar multifidus muscle activation. After that, the subject will be asked to perform 2 repetitions of maximum voluntary isometric contraction (MVIC) of back extensor muscle with 1 minute rest between repetitions. Rater-A will measure right and left lumbar multifidus muscle activation during MVIC and record back extension force from hand-held dynamometer for both repetitions. The data from repetition 1 and 2 will be used to establish intra-rater reliability of ultrasound imaging measurement and calculate minimal detectable change, while data from right and left lumbar multifidus muscles will be used to determine the difference between right and left sides. Subject will be asked to rate the rating of perceived exertion (RPE) and take 5 minute rest to prevent muscle fatigue. After rest period, rater-B will perform exact process as rater-A. These data will be used to establish inter-rater reliability of ultrasound imaging measurement. Rater-A and rater-B are blinded to the subject's group.

The NMES electrodes will be placed on bilateral lumbar multifidus muscles (positive electrode at L3 and negative electrode at L5). Ultrasound transducer will be placed at L4-5 facet joint to capture lumbar multifidus muscle activation. The NMES will be first set at faradic mode (20 Hz, 1 ms). The investigator will increase the intensity at 1 mA increment. Ultrasound imaging data will be recorded, while subject will be asked to rate the 0-10 level of discomfort every 5 mA increment. Rater-A and rater-B will record the intensity used to elicit observable lumbar multifidus muscle contraction. The NMES intensity will increase until maximum level of discomfort (10 out of 10). Subject will be asked to rate the RPE and take a rest period for 10 minutes to prevent muscle fatigue. After rest period, the NMES will be set at interferential mode (6000 Hz, beat frequency 20-50 Hz, scanning effect). The investigator will repeat the entire data collection process. Data from two modes of stimulation will be used to determine the appropriate mode and dose to activate lumbar multifidus muscles.

To determine the feasibility of proposed protocol, the NMES will be set at interferential mode. The investigator will increase NMES intensity until lumbar multifidus muscle 10% increase in thickness. Then, subject will be asked to perform MVIC of back extensor muscle. Rater-A will measure right and left lumbar multifidus muscle activation during MVIC and record back extension force from hand-held dynamometer attached to the thorax. The investigator will decrease NMES intensity to zero. Subject will rest for 10 minutes. After that, the subject will be asked to perform another MVIC of lumbar multifidus muscle without NMES. Rater-A will measure lumbar multifidus muscle activation and record back extension force. The NMES electrodes will be removed and subject's skin will be cleaned. The data (MVIC and MVIC+NMES) will be used to preliminarily determine the existence of arthrogenic muscle inhibition of lumbar multifidus muscle. In addition, the MVIC data without NMES between pre- and post-NMES will be used to determine the existence of retention effect of NMES.

To determine the feasibility of proposed intervention, the NMES will be applied using interferential mode on bilateral lumbar multifidus muscles. The investigator will increase the intensity up to the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total NMES time is 15 minutes. This intervention dose is based on previous studies by Hicks et al. Quadruped rocking exercise will be used as a motor control training in this study. This exercise is based on movement system impairment concept. Subject will be asked to perform quadruped position with spine in neutral position, shoulder and hip in 90 degrees, hips centered over knees, and feet pointing away from body with the dorsum of the feet on the support surface. Then, the subject will be asked to perform rocking back by pushing back with both hands. This verbal instruction will be given to the subject as "Keep your back straight throughout the movement. Think about moving in your hips and not your back. Move in the hips equally". Subject performs rocking back to the position that cause observable and/or palpable posterior pelvic rotation. The subject will be asked to perform rocking back to this target point supervised by the investigator for 10 repetitions followed by 1 minute resting period to minimize muscle fatigue. Subject will be asked to rate the RPE after completion of 10 repetitions. Then, the investigator will re-evaluate the target point again for the next 10 repetitions. This process will be continuously performed for 15 minutes.

After completion of intervention, subject will undergo post-intervention data collection using the same protocol, except only rater-A will perform the post-intervention data collection. The NMES electrodes will be re-applied to bilateral lumbar multifidus muscles. Ultrasound transducer will be re-placed at L4-5 facet joint, and hand-held dynamometer will be re-placed at the thorax. Subject will be asked to perform 2 repetitions of MVIC of back extensor muscle with 1 minute rest between repetitions. Rater-A will measure right and left lumbar multifidus muscle activation during MVIC and record back extension force from hand-held dynamometer for both repetitions. The investigator will increase NMES intensity until lumbar multifidus muscle 10% increase in thickness. Then, subject will be asked to perform MVIC of back extensor muscle. Rater-A will measure right and left lumbar multifidus muscle activation during MVIC and record back extension force from hand-held dynamometer attached to the thorax. The investigator will decrease NMES intensity to zero. Subject will rest for 10 minutes. After that, the subject will be asked to perform another MVIC of lumbar multifidus muscle without NMES. Rater-A will measure lumbar multifidus muscle activation and record back extension force. The NMES electrodes will be removed and subject's skin will be cleaned. Pre- and post-intervention data will be used to determine the feasibility of the proposed intervention.

Phase II: Randomized controlled trial study Phase II study will use a sample of convenience between the ages of 20 and 40. Subjects with and without history of low back pain will be recruited by flyers posted in 2 university physical therapy clinics, as well as word of mouth from subjects and friends. Subjects who are interested in participation will undergo a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If they meet all inclusion criteria, the consent process will be performed.

After obtaining the written informed consent, all subjects will fill out the information sheet for demographic data. Then, subjects will be asked to change their cloth to lab tank top to expose their lower back area. The same body landmarks as preliminary study will be identified. The subjects will be in prone position on treatment table with thorax (T3 level) and pelvis (S2 level) securely fastened to the bed. Hand-held dynamometer will be placed at the thorax to measure back extension force. The NMES electrodes will be placed to bilateral lumbar multifidus muscles, and the system will be set at interferential mode. Then, ultrasound transducer will be placed at right L4-5 facet joint by rater-A.

Subject will be asked to perform 2 repetitions of MVIC of back extensor muscle with 1 minute rest between repetitions. Rater-A will measure right and left lumbar multifidus muscle activation at rest and during MVIC, as well as record back extension force from hand-held dynamometer for both repetitions. The investigator will increase NMES intensity until lumbar multifidus muscle 10% increase in thickness. Then, subject will be asked to perform MVIC of back extensor muscle. Rater-A will measure right and left lumbar multifidus muscle activation during MVIC and record back extension force from hand-held dynamometer attached to the thorax. The NMES electrodes will be removed and subject's skin will be cleaned. The data (MVIC and MVIC+NMES) will be used to determine the existence of arthrogenic muscle inhibition of lumbar multifidus muscle. After pre-intervention data collection, subjects with impaired LPC will be randomly assigned to either combined NMES with motor control training group (COMB), or motor control training alone group (MCT) using randomly generated number in concealed envelopes.

The COMB group will receive the NMES using interferential mode on bilateral lumbar multifidus muscles. The intensity will be set at the subject's maximum tolerance. Stimulation will be set at 10 seconds on and 60 seconds off to minimize muscle fatigue. The total NMES time is 15 minutes. After the NMES, the COMB group will receive 30 minutes motor control training based on movement system impairment concept. This motor control training will focus on the control of the lumbar multifidus muscle in various functional tasks. It is believed to restore the motor units in individuals with arthrogenic muscle inhibition. This motor control training with take approximately 30 minutes. The COMB group will receive intervention twice a week for 8 weeks. We use the 8-week motor training program because several studies have showed significant improvement after 8-week exercise program.1,8 For subjects in MCT group, they will receive placebo NMES (no electrical current) and the same motor control training program as the COMB group. Therapist who provides motor control training will be blinded to the group assignment. After completion of the intervention program, each subject will undergo post-intervention data collection immediately after the first session (Post-1) and after 8-week (Post-2) of intervention to determine the effect of combined neuromuscular electrical stimulation and motor control training in individual with impaired lumbopelvic control.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for individuals without impaired LPC

  1. Between the ages of 20 and 40
  2. No history of LBP that interferes with activities of daily living and/or required treatment
  3. No aberrant movement pattern during active forward bend test
  4. Passive straight leg raising test (SLR) less than 91 degrees
* The inclusion criteria for individuals with impaired LPC

  1. Between the ages of 20 and 40
  2. A recurrent pattern of LBP at least two episodes that interfered with activities of daily living and/or required treatment
  3. Presenting aberrant movement pattern during active forward bend test
  4. Passive straight leg raising test (SLR) greater than 91 degrees

Exclusion Criteria:

1. History of seizure for either the subject or any family member
2. Implanted pacemaker
3. Clinical signs of systemic disease
4. Definitive neurologic signs including pain, weakness or numbness in the lower extremity
5. Previous spinal surgery
6. Diagnosed osteoporosis, severe spinal stenosis, and/or inflammatory joint disease
7. Any lower extremity condition that would potentially alter trunk movement
8. Vestibular dysfunction
9. Extreme psychosocial involvement
10. Body mass index (BMI) greater than 30 kg/m2
11. Active treatment of another medical illness that would preclude participation in any aspect of the study
12. Menstruation or pregnancy (for female subject)
13. Diagnosed herniated nucleus pulposus (HNP)
14. Pain medication usage (e.g., NSAID)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle thickness of lumbar multifidus muscle at baseline. | This outcome will be collected at baseline.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle thickness.
Muscle thickness of lumbar multifidus muscle after the first intervention. | This outcome will be collected at immediately after the first intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle thickness.
Muscle thickness of lumbar multifidus muscle after 8-week intervention. | This outcome will be collected at immediately after 8-week intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle thickness.
Cross-sectional area of lumbar multifidus muscle at baseline. | This outcome will be collected at baseline.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle cross-sectional area.
Cross-sectional area of lumbar multifidus muscle after the first intervention. | This outcome will be collected at immediately after the first intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle cross-sectional area.
Cross-sectional area of lumbar multifidus muscle after 8-week intervention. | This outcome will be collected at immediately after 8-week intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle cross-sectional area.
Pennation angle of lumbar multifidus muscle at baseline. | This outcome will be collected at baseline.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle pennation angle.
Pennation angle of lumbar multifidus muscle after the first intervention. | This outcome will be collected at immediately after the first intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle pennation angle.
Pennation angle of lumbar multifidus muscle after 8-week intervention. | This outcome will be collected at immediately after 8-week intervention.
  The ultrasound imaging device will be used to measure lumbar multifidus muscle pennation angle.

SECONDARY OUTCOMES:
Lumbar and hip muscle length. | This outcome will be collected at baseline only.
  Muscle length will be measured by goniometer using modified Thomas and Ober's tests.
Abdominal and back muscle strength. | This outcome will be collected at baseline only.
  Muscle strength will be measured by hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The IPD of this study will be shared upon official request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The supporting information will be sent upon official request.
Access Criteria: Having an official written request.

REFERENCES:
- [Background] Kiesel KB, Uhl TL, Underwood FB, Rodd DW, Nitz AJ. Measurement of lumbar multifidus muscle contraction with rehabilitative ultrasound imaging. Man Ther. 2007 May;12(2):161-6. doi: 10.1016/j.math.2006.06.011. Epub 2006 Sep 14. PMID 16973400
- [Background] Teyhen D, Koppenhaver S. Rehabilitative ultrasound imaging. J Physiother. 2011;57(3):196. doi: 10.1016/S1836-9553(11)70044-3. PMID 21843838
- [Background] Baek SO, Cho HK, Kim SY, Jones R, Cho YW, Ahn SH. Changes in deep lumbar stabilizing muscle thickness by transcutaneous neuromuscular electrical stimulation in patients with low back pain. J Back Musculoskelet Rehabil. 2017;30(1):121-127. doi: 10.3233/BMR-160723. PMID 27341642
- [Background] Hicks GE, Sions JM, Velasco TO, Manal TJ. Trunk Muscle Training Augmented With Neuromuscular Electrical Stimulation Appears to Improve Function in Older Adults With Chronic Low Back Pain: A Randomized Preliminary Trial. Clin J Pain. 2016 Oct;32(10):898-906. doi: 10.1097/AJP.0000000000000348. PMID 26736024
- [Background] Sung W PT, PhD, Wong A BS, MS, Pourshogi A PhD, Pourrezaei K PhD, Silfies S PT, PhD. Near infrared spectroscopy confirms recruitment of specific lumbar extensors through neuromuscular electrical stimulation. Physiother Theory Pract. 2020 Apr;36(4):516-523. doi: 10.1080/09593985.2018.1488908. Epub 2018 Jun 28. PMID 29952686
- [Derived] Songjaroen S, Sungnak P, Piriyaprasarth P, Wang HK, Laskin JJ, Wattananon P. Combined neuromuscular electrical stimulation with motor control exercise can improve lumbar multifidus activation in individuals with recurrent low back pain. Sci Rep. 2021 Jul 20;11(1):14815. doi: 10.1038/s41598-021-94402-2. PMID 34285318